CLINICAL TRIAL: NCT04689789
Title: The Role of Quantitative Deep Capillary Plexus in the Pathogenesis of Retinal Angiomatous Proliferation: an Optical Coherence Tomography Angiography Study.
Brief Title: OCTA and Retinal Angiomatous Proliferation
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 2912/20
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with RAP: Patients with previous diagnosis of retinal angiomatous proliferation
  Interventions: Diagnostic Test: optical coherence tomography angiography
- Patients with reticular pseudodrusen: Patients with previous diagnosis of reticular pseudodrusen
  Interventions: Diagnostic Test: optical coherence tomography angiography
- Control group: Healthy eyes without actual and previous ocular diseases
  Interventions: Diagnostic Test: optical coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: optical coherence tomography angiography — optical coherence tomography aniography is a non-invasive, fast, diagnostic imaging technique that evaluates the retinal vascular network

SUMMARY:
To investigate, using optical coherence tomography angiography, the retinal vascular features in patients affected by RAP.

DETAILED DESCRIPTION:
Retinal vascular anomalous complex represents a distinct form of neovascularization in patients with age-related macular degeneration.

The study investigated the changes in retinal vascular network using optical coherence tomography angiography, a novel and non invasive diagnostic technique that allows to better understand the pathophysiologic mechanism of this neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* age older than 65 years
* diagnosis of retinal angiomatous proliferation and reticular pseudodrusen
* absence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* absence of significant lens opacities, low-quality OCT-A images.

Exclusion Criteria:

* age older than 80 years
* absence of diagnosis of retinal angiomatous proliferation and reticular pseudodrusen
* presence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* presence of significant lens opacities, low-quality OCT-A images.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The participans were older than 65 years with diagnosis of age-related macular degeneration and in particular retinal angiomatous proliferation and reticular pseudodrusen.
  They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal vascular network in patients with age-related macular degeneration, using optical coherence tomography angiography, compared to controls | 15 months
  The parameters analyzed by optical coherence tomography angiography were: vessel density of superficial capillary plexus and deep capillary plexus

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Naples, Napoli, Italy